CLINICAL TRIAL: NCT03900169
Title: Familial Hypercoleresremia as Risk Factor in Stemi Patient Underwent Ppci
Brief Title: Familial Hypercolerstremia as Risk Factor in Stemi Patient Who Underwent Ppci
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Harby, Principle investigator, Assiut University
Other Study IDs: Familial hypercolerstremia
Record Dates: First submitted 2019-03-25; First posted 2019-04-02 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stemi patient: Stemi patient who underwent Ppci
  Interventions: Genetic: Genetic

INTERVENTIONS:
Genetic: Genetic — Lipid profile

SUMMARY:
Famulial hypercolerstremia as risk factor

DETAILED DESCRIPTION:
Familial hypercolerestremia ad risk factor in stemi patient who underwent Ppci

ELIGIBILITY:
Inclusion Criteria:

-all patient that underwent Ppci

Exclusion Criteria:

* Previous ischemic patient
* Patient with raised renal chemistry
* Patient for CABG

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Stemi patient
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between familial hypercolerstremia and prognosis of patients in PPCI | One year
  Correlation between familial hypercolerstremia and prognosis of patients in PPCI
Correlation between non familial hypercolerstremia and prognosis of patients in PPCI | One year
  Correlation between non familial hypercolerstremia and prognosis of patients in PPCI

CONTACTS AND LOCATIONS:
Locations (1):
- Amira harby, Asyut, Egypt